CLINICAL TRIAL: NCT03453541
Title: A Randomized, Double-blinded, Placebo-controlled Study of Ketorolac Use in Pediatric Patients Undergoing Tonsillectomy
Brief Title: Ketorolac Use in Pediatric Patients Undergoing Tonsillectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited recruitment resources.
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Farzana Afroze, Assistant Professor of Anesthesiology, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4923
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2021-09

CONDITIONS: Analgesic Adverse Reaction
MeSH Terms: interventions — Ketorolac Tromethamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: CRNAs, PACU nurses, and participants are all blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac Tromethamine (Experimental): This group receives Ketorolac Tromethamine 0.5 mg/kg IV up to a maximum dose of 30mg, in the form of Ketorolac Tromethamine solution for IV/IM use 30mg/ml single dose vial at the completion of the tonsillectomy in the operating room.
  Interventions: Drug: Ketorolac Tromethamine
- 0.9% Normal Saline (Placebo Comparator): This group will receive 0.9% Normal Saline solution 1ml/60kg up to 1ml IV bolus (an equivalent volume as per kg Ketorolac Tromethamine dose) at the completion of the tonsillectomy in the operating room.
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Ketorolac Tromethamine 0.5 mg/kg IV up to a maximum dose of 30mg, in the form of Ketorolac Tromethamine solution for IV/IM use 30mg/ml single dose vial at the completion of the tonsillectomy in the operating room.
  Other Names: Toradol
  Arms: Ketorolac Tromethamine
Drug: 0.9% Normal Saline — 0.9 % Normal saline 1ml/60kg up to a maximum dose of 1ml IV bolus (an equivalent volume as per kg Ketorolac Trimethamine dose) at the completion of the tonsillectomy in the operating room.
  Other Names: 0.9% Sodium Chloride
  Arms: 0.9% Normal Saline

SUMMARY:
This prospective, randomized, double blinded study is designed to compare the bleeding rates of ketorolac vs. placebo when used for post tonsillectomy pain control in pediatric patients ages 2-18.

DETAILED DESCRIPTION:
Tonsillectomy/adenoidectomy is an elective operation, mainly in the pediatric population. This procedure is performed by Dr. Jason Mouzakes and the otolaryngology residents under his supervision. The location of the research is at the Albany Medical Center Hospital, Main Campus and South Clinical Campus. Duration of this study for each individual patient will be set at 14 days post procedure, taking into account that bleeding risk with this procedure is highest within the first 2 weeks post-operatively. Data will be obtained within 90 days after discharge from the hospital by telephone interview with the parents or hospital record. The investigators plan to enroll at least 600 patients, 300 in each group, ASA physical status I to III and age 2 years to 18 years old (inclusive). Parents and children may be informed about the study at the time when surgery is planned during initial office visit. Enrollment in the study will be done on the day of the surgery, after the Anesthesiologist or Otolaryngology/Anesthesiology Resident explains the purpose, benefits and possible risks of the study and answers all questions of the parents. Before enrollment is finalized, informed consent and informed assent, if applicable, to take part in a human research study will be obtained.

At the completion of surgery, patients will be transferred to the post-anesthesia care unit (PACU). Additional pain medication if needed in the PACU will be acetaminophen 15mg/kg oral solution or opioid medications at discretion of treating anesthesiologist. Acetaminophen will only be given in PACU if it was not received pre-operatively. Patients will be discharged to home from the PACU or 2nd level short-stay recovery unit (at South Clinical Campus) when standard criteria are met for each patient per protocol.

Randomization Plan:

Patients will be randomized by a card system. There will be 600 cards with 300 labeled (K) for ketorolac group and 300 labeled (NS) for placebo group along with the assigned subject number. Preservative free 0.9% normal saline will be used as placebo. Randomization will be done using www.randomization.com which will generate a randomization sequence with a concealed blocking schedule. A non-investigator will prepare envelopes numbered sequentially, each containing a card indicating the subject number (sequentially numbered 1 - 600) and group as randomized by above plan. Envelopes are opened only upon obtaining consent maintaining allocation concealment until treatment is initiated. Patients are therefore assigned a subject number at the initiation of the study. The non-treating anesthesiologist will open the next sequential envelope (starting from envelope #1) and draw up the specified drug and give the drug with a patient label to the treating anesthesiologist. The non-treating anesthesiologist will also tell the treating anesthesiologist the patient's subject number so it may be recorded on the individual data collection sheet. The non-treating anesthesiologist will place a patient label on the drug card and store the card in the anesthesiology office, specifically Dr Afroze's office inside of room D108. Dr Afroze's office is locked and has minimal access. The patient drug cards will be accessed by the research team two weeks after the surgery date to record patient data.

The PACU nurses, surgeon, residents, and treating anesthesiologist will all be blinded and may perform the PACU scoring and data collection. Study drugs will be documented the same exact way on the anesthesia records for all the study patients. All the study patients' charts will have both drugs documented as IN study drug dose in mg. The doses of the drugs are pre-calculated based on the patient's weight and will be drawn by a non-treating anesthesiologist and administered by the treating anesthesiologist at the time of the surgery.

Patients for our study will be recruited from the Pediatric ENT clinical practice of Dr. Mouzakes. Surgery, anesthesia, and postoperative recovery will take place at the Albany Medical Center Hospital, Main Campus and South Clinical Campus. The investigators plan to enroll 600 children, age of 2 to 18 years old (inclusive) and ASA physical status I to III. The investigators anticipate completing our study in 12 to 24 months.

This study will have power of 81% to show that the bleeding rate for new treatment (ketorolac) is at least as low as the event rate for the control group. This assumes that the true event rates for the active control and new treatment populations are precisely equal (at 2.0%), that a difference of 3.0% or less is unimportant, that the sample size in the two groups will be 280 and 280, and that alpha (1 tailed) is set at .05.

Formally, the null hypothesis is that the event rate for new treatment is 3.0 percentage points higher than the event rate for active control, and the study has power of 81.3% to reject this null. Equivalently, the likelihood is 81.3% that the 95.0% confidence interval for the difference in event rates will exclude a 3.0 point difference in favor of active control.

The primary endpoint, bleeding rates, will be compared between the two groups by Chi-square test (or Fisher's exact test if expected values are 5 or less). Other secondary categorical data (readmission, PACU nausea/vomitting) will be analyzed similarly. Continuous data (opioid administrations, PACU pain scores, length of stay in recovery units) will be compared with an independent sample t-test or Mann-Whitney test if data demonstrates significant non-normality. Multivariable analysis will be used to determine if bleeding is associated with the covariates age, gender, weight, ASA status, and primary or secondary diagnoses.

The risks of the study include the risks of possible allergic reactions to ketorolac in patients with no previously known drugs allergies, and possible decreased pain control for some patients. However, as is standard of practice, all patients with uncontrolled post-operative pain will have additional acetaminophen or opioid medications administered as needed for pain in the post-operative units under the guidance of the treating anesthesiologist. As previously demonstrated, ketorolac intravenous & intramuscular have been shown in the anesthesiology literature to be safe with a low incidence of side effects. Patient's parents will be informed of other possible side effects of ketorolac including platelet dysfunction with prolonged bleeding at operative site, gastrointestinal bleeding, and renal dysfunction. There are no described long term side effects from single intraoperative application of ketorolac. Side-effects that have been noticed in other studies are minimal and transient. Patient's parents will have access to the investigator and ER department 24 hours a day, 7 days a week if any concerns appear.

The major benefit from IV ketorolac for patients is potential of adequate pain control for tonsillectomy with decreased use of opioid analgesia, ameliorating possible negative side effects of narcotics such as respiratory depression and nausea/vomiting. Achieving adequate pain control in tonsillectomy patients leads to improved oral intake and decreased risk of dehydration. Additionally, results of this study will be contributing to improvement in pain management for future patients undergoing tonsillectomy surgery. Overall, The investigators feel that the risks involved with this study are minimal and potential benefits are quite large.

The PHI to be collected includes the medical record number and date of birth to identify the range of age of the participants, possible allergy to medications, and brief past medical history relevant to the study.

If consent is not obtained, the patient will not be included in the study and will receive standard assessment and care, which typically includes single dose 0.5mg/ kg ketorolac at the completion of the procedure and additional pain medications in recovery areas as needed, such as acetaminophen or opioids. At any point in the study, the subject may choose to discontinue participation and opt for standard treatment.

ELIGIBILITY:
Inclusion Criteria:

-ASA physical status I to III, age of 2 years to 18 years old (inclusive) scheduled for elective tonsillectomy with or without adenoidectomy.

Exclusion Criteria:

-Exclusion criteria are: allergy to any nonsteroidal anti-inflammatory medications, bleeding disorders, history of gastrointestinal bleeding, renal impairment, severe asthma, cardiac/hepatic disease, use of anticoagulation, recent NSAID use (within last 72 hours) or any other medical problem that in the opinion of investigator would interfere with study participation.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Rebleeding rate requiring operative intervention | 2 weeks post-operative
  Rebleeding rate requiring operative intervention measured by recording either yes or no the patient did or did not returned to the OR for bleeding related to recent tonsillectomy. Requiring operative intervention would be a worse outcome than not requiring operative intervention.

SECONDARY OUTCOMES:
PACU length of stay | Immediately after operation
  PACU length of stay in minutes from admission to discharge. The longer the length of PACU stay the worse the outcome.
Post-operative opioid dosage | Immediately after operation
  Post- operative opioid requirement in mg of Morphine/ Morphine equivalent. The greater the amount of opioid used the worse the outcome.
Post-operative pain score | Immediately after operation
  Pain scores ranging from 0 to 5 will be collected using the Visual Analogue Pain. scale. A score of 0 indicates no pain and a score of 5 indicates unbearable pain. The greater the pain score would indicate a worse outcome.
Presence of post-operative nausea/vomiting | Immediately after operation
  The presence of post operative nausea or vomiting while in the PACA measured by either yes or no. The presence of pots-operative nausea or vomiting would indicate a worse outcome.
Number of emergency room visits/admissions | 2 weeks post-operative
  The number of actual emergency room visits by the patient measured numerically from 1 to infinity. The greater the number of emergency room visits would indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Farzana Afroze, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Chan DK, Parikh SR. Perioperative ketorolac increases post-tonsillectomy hemorrhage in adults but not children. Laryngoscope. 2014 Aug;124(8):1789-93. doi: 10.1002/lary.24555. Epub 2014 May 27. PMID 24338331
- [Background] Riggin L, Ramakrishna J, Sommer DD, Koren G. A 2013 updated systematic review & meta-analysis of 36 randomized controlled trials; no apparent effects of non steroidal anti-inflammatory agents on the risk of bleeding after tonsillectomy. Clin Otolaryngol. 2013 Apr;38(2):115-29. doi: 10.1111/coa.12106. PMID 23448586
- [Background] Lee WT, Witsell DL, Parham K, Shin JJ, Chapurin N, Pynnonen MA, Langman A, Nguyen-Huynh A, Ryan SE, Vambutas A, Roberts RS, Schulz K. Tonsillectomy Bleed Rates across the CHEER Practice Research Network: Pursuing Guideline Adherence and Quality Improvement. Otolaryngol Head Neck Surg. 2016 Jul;155(1):28-32. doi: 10.1177/0194599816630523. PMID 27371623
- [Background] Windfuhr JP, Chen YS, Remmert S. Hemorrhage following tonsillectomy and adenoidectomy in 15,218 patients. Otolaryngol Head Neck Surg. 2005 Feb;132(2):281-6. doi: 10.1016/j.otohns.2004.09.007. PMID 15692542
- [Background] Lane JC, Dworkin-Valenti J, Chiodo L, Haupert M. Postoperative tonsillectomy bleeding complications in children: A comparison of three surgical techniques. Int J Pediatr Otorhinolaryngol. 2016 Sep;88:184-8. doi: 10.1016/j.ijporl.2016.07.007. Epub 2016 Jul 11. PMID 27497410
- [Background] Bailey R, Sinha C, Burgess LP. Ketorolac tromethamine and hemorrhage in tonsillectomy: a prospective, randomized, double-blind study. Laryngoscope. 1997 Feb;107(2):166-9. doi: 10.1097/00005537-199702000-00006. PMID 9023238
- [Background] Judkins JH, Dray TG, Hubbell RN. Intraoperative ketorolac and posttonsillectomy bleeding. Arch Otolaryngol Head Neck Surg. 1996 Sep;122(9):937-40. doi: 10.1001/archotol.1996.01890210017004. PMID 8797556
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Background] Moodie JE, Brown CR, Bisley EJ, Weber HU, Bynum L. The safety and analgesic efficacy of intranasal ketorolac in patients with postoperative pain. Anesth Analg. 2008 Dec;107(6):2025-31. doi: 10.1213/ane.0b013e318188b736. PMID 19020154
- [Background] Ketorolac., Drug Facts and Comparisons 4.0 (online). I. Wolters Kluwer Health, Editor. 2011.
- [Background] Ketorolac. National Cancer Institute Drug Dictionary.
- [Background] Gupta A, Daggett C, Ludwick J, Wells W, Lewis A. Ketorolac after congenital heart surgery: does it increase the risk of significant bleeding complications? Paediatr Anaesth. 2005 Feb;15(2):139-42. doi: 10.1111/j.1460-9592.2005.01409.x. PMID 15675931
- [Background] Aldrink JH, Ma M, Wang W, Caniano DA, Wispe J, Puthoff T. Safety of ketorolac in surgical neonates and infants 0 to 3 months old. J Pediatr Surg. 2011 Jun;46(6):1081-5. doi: 10.1016/j.jpedsurg.2011.03.031. PMID 21683202
- [Background] Papacci P, De Francisci G, Iacobucci T, Giannantonio C, De Carolis MP, Zecca E, Romagnoli C. Use of intravenous ketorolac in the neonate and premature babies. Paediatr Anaesth. 2004 Jun;14(6):487-92. doi: 10.1111/j.1460-9592.2004.01250.x. PMID 15153212
- [Background] Lynn AM, Bradford H, Kantor ED, Andrew M, Vicini P, Anderson GD. Ketorolac tromethamine: stereo-specific pharmacokinetics and single-dose use in postoperative infants aged 2-6 months. Paediatr Anaesth. 2011 Mar;21(3):325-34. doi: 10.1111/j.1460-9592.2010.03484.x. Epub 2010 Dec 29. PMID 21199130
- [Background] Cohen MN, Christians U, Henthorn T, Vu Tran Z, Moll V, Zuk J, Galinkin J. Pharmacokinetics of single-dose intravenous ketorolac in infants aged 2-11 months. Anesth Analg. 2011 Mar;112(3):655-60. doi: 10.1213/ANE.0b013e3182075d04. Epub 2011 Jan 13. PMID 21233498
- [Background] Pappas AL, Fluder EM, Creech S, Hotaling A, Park A. Postoperative analgesia in children undergoing myringotomy and placement equalization tubes in ambulatory surgery. Anesth Analg. 2003 Jun;96(6):1621-1624. doi: 10.1213/01.ANE.0000064206.51296.1D. PMID 12760984
- [Background] Zuppa AF, Mondick JT, Davis L, Cohen D. Population pharmacokinetics of ketorolac in neonates and young infants. Am J Ther. 2009 Mar-Apr;16(2):143-6. doi: 10.1097/MJT.0b013e31818071df. PMID 19300040
- [Background] Neri E, Maestro A, Minen F, Montico M, Ronfani L, Zanon D, Favret A, Messi G, Barbi E. Sublingual ketorolac versus sublingual tramadol for moderate to severe post-traumatic bone pain in children: a double-blind, randomised, controlled trial. Arch Dis Child. 2013 Sep;98(9):721-4. doi: 10.1136/archdischild-2012-303527. Epub 2013 May 23. PMID 23702435
- [Background] Gupta A, Daggett C, Drant S, Rivero N, Lewis A. Prospective randomized trial of ketorolac after congenital heart surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):454-7. doi: 10.1053/j.jvca.2004.05.024. PMID 15365927
- [Background] Perez-Urizar J, Aguilar-Cota ME, Herrera JE, Flores-Murrieta FJ. Comparative bioavailability of ketorolac tromethamine after intramuscular and sublingual administration. Proc West Pharmacol Soc. 2002;45:6-7. No abstract available. PMID 12434509
- [Background] Drover DR, Hammer GB, Anderson BJ. The pharmacokinetics of ketorolac after single postoperative intranasal administration in adolescent patients. Anesth Analg. 2012 Jun;114(6):1270-6. doi: 10.1213/ANE.0b013e31824f92c2. Epub 2012 Mar 30. PMID 22467894
- [Background] Lieh-Lai MW, Kauffman RE, Uy HG, Danjin M, Simpson PM. A randomized comparison of ketorolac tromethamine and morphine for postoperative analgesia in critically ill children. Crit Care Med. 1999 Dec;27(12):2786-91. doi: 10.1097/00003246-199912000-00030. PMID 10628627
- [Background] Forrest JB, Heitlinger EL, Revell S. Ketorolac for postoperative pain management in children. Drug Saf. 1997 May;16(5):309-29. doi: 10.2165/00002018-199716050-00003. PMID 9187531
- [Background] 26. Ketorolac: Peds Dosing. 2017: Epocrates.
- [Background] 27. Ketorolac Dosage. Drugs.com.
- [Background] Lynn AM, Bradford H, Kantor ED, Seng KY, Salinger DH, Chen J, Ellenbogen RG, Vicini P, Anderson GD. Postoperative ketorolac tromethamine use in infants aged 6-18 months: the effect on morphine usage, safety assessment, and stereo-specific pharmacokinetics. Anesth Analg. 2007 May;104(5):1040-51, tables of contents. doi: 10.1213/01.ane.0000260320.60867.6c. PMID 17456651
- [Background] Liu Y, Seipel C, Lopez ME, Nuchtern JG, Brandt ML, Fallon SC, Manyang PA, Tjia IM, Baijal RG, Watcha MF. A retrospective study of multimodal analgesic treatment after laparoscopic appendectomy in children. Paediatr Anaesth. 2013 Dec;23(12):1187-92. doi: 10.1111/pan.12271. Epub 2013 Sep 25. PMID 24112856